CLINICAL TRIAL: NCT04203901
Title: A Phase 2b Randomized Trial of Autologous Dendritic Cell Immunotherapy (CMN-001) Plus Standard Treatment of Advanced Renal Cell Carcinoma
Brief Title: Dendritic Cell Immunotherapy Plus Standard Treatment of Advanced Renal Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic corporate decision
Sponsor: CoImmune (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMN-001-1
Record Dates: First submitted 2019-12-10; First posted 2019-12-18 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-09

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Combination Arm (Experimental): CMN-001 dosing (1x10^7 DC/dose) is initiated at Visit 2 during 1st line therapy and through 2nd line therapy. CMN-001 is administered as 1 dose every 3 weeks for 3 doses (Induction phase), followed by maintenance doses, 1 every 4 weeks for 7 doses (Maintenance phase), followed by booster doses, 1 dose every 12 weeks (Booster phase). 1st line therapy, Nivolumab (3mg/kg) + Ipilimumab (1 mg/kg) will be administered at 3 week intervals for 4 administrations starting at visit 1. Followed by Nivolumab (3 mg/kg) administration every 4 weeks until progression. After progression, 2nd line therapy with lenvatinib (18mg/day) + everolimus (5mg/day) until discontinuation criteria are met.
  Interventions: Biological: CMN-001; Biological: Nivolumab+Ipilimumab; Drug: Lenvatinib+Everolimus
- Standard Treatment (Active Comparator): 1st line therapy, Nivolumab (3mg/kg) + Ipilimumab (1 mg/kg) will be administered at 3 week intervals for 4 administrations starting at visit 1. Followed by Nivolumab (3 mg/kg) administration every 4 weeks until progression. After progression 2nd line therapy with lenvatinib (18mg/day) + everolimus (5mg/day) until discontinuation criteria are met.
  Interventions: Biological: Nivolumab+Ipilimumab; Drug: Lenvatinib+Everolimus

INTERVENTIONS:
Biological: CMN-001 — Autologous Dendritic Cell Therapy
  Arms: Combination Arm
Biological: Nivolumab+Ipilimumab — anti-PD-1 and anti-CTLA4 antibodies
Drug: Lenvatinib+Everolimus — TKI+mTOR inhibitors

SUMMARY:
CMN-001 is an autologous, tumor antigen-loaded dendritic cell immunotherapy. The active components of CMN-001 are autologous, matured dendritic cells, which have been co-electroporated with both in vitro transcribed (IVT) RNA from an autologous tumor specimen and CD40L RNA. CMN-001 is indicated for treatment of intermediate/poor risk patients with advanced renal cell carcinoma (RCC) in combination with nivolumab plus ipilimumab as first line therapy and in combination with lenvatinib plus everolimus as 2nd line therapy post 1st line failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Advanced disease histologically assessed as RCC, with predominantly clear cell histology
3. Metastatic disease (measurable or non-measurable) that can be monitored throughout the course of study participation per iRECIST
4. Subjects who are candidates for standard first-line therapy
5. Time from initial RCC diagnosis to initiation of systemic treatment (Nivolumab+Ipilimumab) of <1 year
6. Karnofsky Performance Status (KPS) ≥ 70%
7. Resolution of all acute toxic effects of prior radiotherapy or surgical procedures to Grade ≤ 1 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
8. Adequate hematologic function, as defined by central laboratory values for all three of the following criteria:

   1. Absolute neutrophil count (ANC) LLN, and
   2. Platelets 75,000/mm3 or 75.0 x 109/L, and
   3. Hemoglobin (Hgb) 8.0 g/dL
9. Adequate renal function, as defined by either of the following criteria:

   1. Serum creatinine 1.5 x upper limit of normal (ULN),
   2. OR, if serum creatinine greater than 1.5 x ULN, estimated glomerular filtration rate (eGFR) 30 mL/min
10. Adequate hepatic function, as defined by both of the following:

    1. Total serum bilirubin 1.5 x ULN
    2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) 2.5 x ULN or, AST and ALT 5 x ULN if liver function abnormalities are due to underlying malignancy
11. Adequate coagulation function as defined by either of the following criteria:

    1. INR < 1.5 x ULN
    2. For subjects receiving warfarin or LMWH, the subjects must, in the investigator's opinion, be clinically stable with no evidence of active bleeding while receiving anticoagulant therapy. The INR for these patients may exceed 1.5 x ULN if that is the goal of anticoagulant therapy.
12. Negative serum pregnancy test for female subjects with reproductive potential, and agreement of all male and female subjects of reproductive potential to use a reliable form of contraception during the study and for 12 weeks after the last dose of study drug
13. Normal ECG or clinically non-significant finding(s) at Screening, in the Investigator's opinion
14. Able to abstain from taking prohibited drugs, either prescription or non-prescription, during the treatment phase of the study
15. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
16. Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Prior history of malignancy within the preceding 3 years, except for adequately treated in situ carcinomas or non-melanoma skin cancer, adequately treated early stage breast cancer, superficial bladder cancer, and non-metastatic prostate cancer with a normal PSA.
2. History of or known brain metastases, spinal cord compression, or carcinomatous meningitis, or evidence of brain or leptomeningeal disease
3. Patients will be excluded if they have <2 of the following risk factors at Screening:

   1. Time from diagnosis to systemic treatment < 1 year
   2. Hgb < LLN
   3. Corrected calcium > 10.0 mg/dL
   4. KPS < 80%
   5. Neutrophils > ULN
   6. Platelets > ULN
4. NCI CTCAE Grade 3 hemorrhage < 28 days before Visit 1 (Week 0)
5. Clinically significant cardiovascular conditions within 3 months prior to Randomization, which in the Investigator's opinion prohibits the initiation of standard targeted therapy, initiating with sunitinib, including:

   1. Cardiac angioplasty
   2. Myocardial infarction
   3. Unstable angina
   4. Coronary artery by-pass graft or stenting
   5. Class III or IV congestive heart failure (CHF), per NYHA Classification NOTE: Patients with left ventricular ejection fraction (LVEF) < LLN as assessed by either echocardiography or multiple gated acquisition (MUGA) scan, who are asymptomatic and are NOT classified as having NYHA Class III or IV CHF, may be eligible but should be monitored for LVEF changes while on sunitinib therapy as recommended in the current sunitinib prescribing information.
   6. Symptomatic peripheral vascular disease
   7. Cerebrovascular accident (CVA) or transient ischemic attack (TIA)
   8. Symptomatic or uncontrolled pulmonary embolism or deep vein thrombosis (DVT)
   9. Uncontrolled cardiac dysrhythmias of NCI CTCAE Grade ≥ 2, or prolongation of the QTc for males > 450 msec and for females > 470 msec as corrected by either the Fridericia or Bazett formula
   10. Uncontrolled or untreated atrial fibrillation
   11. Poorly controlled hypertension, defined as a systolic blood pressure (SBP), ≥ 150 mm Hg or diastolic blood pressure (DBP) ≥ 90 mm Hg NOTE: Initiation of antihypertensive medication(s) is permitted prior to study entry. Blood pressure must be re-assessed on 2 occasions separated by at least 1 hour. Mean SBP/DBP values must be less than 150/90 for eligibility.
   12. Evidence of active bleeding or a bleeding diathesis at Screening
6. Significant gastrointestinal abnormalities:

   1. Any history of major resection of the stomach or small bowel with ongoing impaired healing.
   2. Malabsorption syndrome with active symptoms in the Investigator's opinion, within 3 months prior to Randomization
   3. Active peptic ulcer, which cannot be appropriately managed in the Investigator's opinion, within 3 months prior to Randomization
   4. Intra-luminal bleeding lesions within 3 months prior to Randomization
   5. History of abdominal fistula or intra-abdominal abscess within 3 months prior to Randomization
7. Pre-existing thyroid abnormality with thyroid function that cannot be appropriately managed with medication, in the Investigator's opinion.
8. Active autoimmune disease or condition requiring chronic immunosuppressive therapy, such as rheumatoid arthritis, systemic lupus erythematous, multiple sclerosis, organ transplant recipient, etc.

   NOTE: Abnormal laboratory values for autoimmunity markers in the absence of other signs/symptoms of autoimmune disease are not exclusionary.
9. Clinically significant infections, including human immunodeficiency virus (HIV), syphilis, and active hepatitis B or C
10. Current treatment with an investigational therapy on another clinical trial
11. Pregnancy or breastfeeding
12. Any serious medical condition or illness considered by the investigator to constitute an unwarranted high risk for investigational treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Through study completion, an average of 2 years
  Patients will be followed for OS until the completion of the study.

SECONDARY OUTCOMES:
Monitor treatment emergent adverse events between both arms | Through study completion, an average of 2 years
  Compare adverse events between both arms
Progression free survival | Through study completion, an average of 2 years
  Progression-free survival from the date of subject randomization as assessed by the investigator per iRECIST.
  Radiological evidence of progression will be derived from tumor imaging assessments at baseline (Screening, Week 0) and restaging scans at Week 13, 21, 29, 37 then every 12 weeks until progression or study withdrawal.
Tumor Response | Through study completion, an average of 2 years
  To compare tumor responses based on iRECIST between study arms

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - SUNY Upstate Medical University, Syracuse, New York
  - Westchester Medical Center, Valhalla, New York
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Houston Methodist, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - West Virginia University Cancer Institute, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No